CLINICAL TRIAL: NCT01801579
Title: Reproducibility of the Ankle-Brachial Index Measurements After a Maximal Exercise
Brief Title: Reproducibility of Ankle Brachial Index After Maximal Exercise
Acronym: RICATEM
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Institut de formation en éducation physique et en sport d'Angers/Les Ponts de Cé (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2012-A01036-37
Record Dates: First submitted 2013-02-18; First posted 2013-03-01 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Normal Subjects
Keywords: Ankle Brachial Index; Maximal exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hemodynamic changes in the lower limbs are very important and rapid after maximal exercise. The automatic method allows a fastest measurement of the Ankle-Brachial Index (ABI). Thus, it appears important to know whether automatic assessment of ABI is as reliable and reproducible as the manual method.

DETAILED DESCRIPTION:
Two methods are mainly used to determine the blood pressure at rest, in a non-invasive way, in order to calculate the Ankle-Brachial Index (ABI). The first method, using a manual sphygmomanometer coupled with a Doppler probe, is considered as the reference method. The second method requires at least one automatic sphygmomanometer. Data from the literature show that these two methods are reproducible to assess ABI at rest. Some authors have reported a better reproducibility of measurements with automatic tool. Others consider that the current accuracy of automatic measurement is insufficient to replace the reference method Doppler. Thus, the aime of the present study is to evaluate whether automatic assessment of ABI is as reliable and reproducible as the manual method.

ELIGIBILITY:
Inclusion Criteria:

* Participant between 18 and 40 years old
* Informed consent signed
* Exclusion Criteria:
* Do not want to participate to the protocol
* Pregnant woman
* Adults to enhanced protection, deprived of their liberty by judicial or administrative authority, without consent hospitalized or admitted to a health facility or social purposes other than research
* Being in a period of exclusion from another biomedical study
* Amputee or with a member dysgenesis
* Not allowed to perform a maximal exercise

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: health volunteers over 18 years old
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Test-retest difference in ankle to brachial pressure index | up to 2 week
  Comparison of differendces observed on test-retest measures with manual and automatic measurements

SECONDARY OUTCOMES:
Duration of recordings. | up to 2 weeks
  Comaprison of the time needed to complete the recording with automatic vs. manual techniques

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BRUNEAU, MD, Principal Investigator — University Hospital, Angers
Locations (1):
- University Hospital, Angers, France